CLINICAL TRIAL: NCT00875784
Title: An Open-label, Randomized, 3-period Crossover Study to Evaluate Sumatriptan Pharmacokinetics for a TREXIMA™ (Sumatriptan Succinate / Naproxen Sodium) Tablet Followed by IMITREX® (Sumatriptan Succinate) Injection 4mg Administered Using the IMITREX STATdose System® and a TREXIMA Tablet Followed by IMI
Brief Title: An Open-label, Randomized, 3-period Crossover Study to Evaluate Sumatriptan Pharmacokinetics for a TREXIMA™ (Sumatriptan Succinate / Naproxen Sodium) Tablet Followed by IMITREX® (Sumatriptan Succinate)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 103629
Record Dates: First submitted 2009-03-26; First posted 2009-04-03 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Migraine Disorders
Keywords: Sumatriptan exposure
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TREXIMA tablet followed by IMITREX injection (4mg) (Experimental): TREXIMA™ (sumatriptan succinate / naproxen sodium) Tablet followed by IMITREX® (sumatriptan succinate) Injection 4mg administered using the IMITREX STATdose System®
  Interventions: Drug: TREXIMA™; Drug: IMITREX® (4mg)
- TREXIMA tablet followed by IMITREX injection (6mg) (Experimental): TREXIMA tablet followed by IMITREX® (sumatriptan succinate) Injection 6mg administered using the IMITREX STATdose System®
  Interventions: Drug: TREXIMA™; Drug: IMITREX® (6mg)
- IMITREX tablet (100mg) (Active Comparator): IMITREX 100mg tablet followed 2 hours later by a second IMITREX 100mg tablet
  Interventions: Drug: IMITREX Tablet 100mg

INTERVENTIONS:
Drug: TREXIMA™ — sumatriptan succinate / naproxen sodium tablet
  Arms: TREXIMA tablet followed by IMITREX injection (4mg); TREXIMA tablet followed by IMITREX injection (6mg)
Drug: IMITREX® (4mg) — sumatriptan succinate injection (4mg) administered using the IMITREX STATdose System®
  Arms: TREXIMA tablet followed by IMITREX injection (4mg)
Drug: IMITREX® (6mg) — sumatriptan succinate injection (6mg) administered using the IMITREX STATdose System®
  Arms: TREXIMA tablet followed by IMITREX injection (6mg)
Drug: IMITREX Tablet 100mg — IMITREX 100mg tablet followed 2 hours later by a second IMITREX 100mg tablet
  Arms: IMITREX tablet (100mg)

SUMMARY:
This study will evaluate the exposure of sumatriptan after administration of TREXIMA (sumatriptan 85mg/naproxen sodium 500mg) followed by a subcutaneous IMITREX injection (4mg or 6mg) 2 hours later compared to administration of a IMITREX 100mg tablet followed by a IMITREX 100mg tablet 2 hours later.

DETAILED DESCRIPTION:
An open-label, randomized, 3-period crossover study to evaluate sumatriptan pharmacokinetics for a TREXIMA™ (sumatriptan succinate / naproxen sodium) Tablet followed by IMITREX® (sumatriptan succinate) Injection 4mg administered using the IMITREX STATdose System® and a TREXIMA tablet followed by IMITREX® (sumatriptan succinate) Injection 6mg administered using the IMITREX STATdose System® compared with an IMITREX Tablet 100mg followed by an IMITREX Tablet 100mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females between 18 and 55 years of age, inclusive. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory studies and other tests.
* Female subjects of non-childbearing potential
* Any subject taking oral contraceptives has been on a stable regimen for at least 2 months prior to screening.
* BMI: 20-30 kg/m2, inclusive.
* Subject is willing and able to provide written informed consent.

Exclusion Criteria:

* Subjects who suffer from migraine attacks.
* Subject has confirmed or suspected ischemic heart disease; angina pectoris, history of myocardial infarction, documented silent ischemia, Prinzmetal's angina-coronary vasospasm, signs, or symptoms consistent with any of the above.
* Subject has evidence or history of ischemic abdominal syndromes, peripheral vascular disease or Raynaud's syndrome.
* Subject has cardiac arrhythmias requiring medication or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
* Subject has a history of cerebrovascular pathology including stroke and/or transient ischemic attacks.
* Subject has a history of congenital heart disease.
* Subject has hypertension at screening.
* Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease.
* Subject has a history of epilepsy or structural brain lesions which lower the convulsive threshold or treated with an antiepileptic drug for seizure control within 5 years prior to screening.
* History of impaired hepatic or renal function.
* Subject is currently taking or has taken in the previous 4 weeks, herbal preparations containing St. John's Wort.
* Use of other prescription or non-prescription drugs, vitamins, herbal and dietary supplements, within 7 days prior to the first dose of study medication.

Note: Excluded from this list are: acetaminophen at doses of less than or equal to 2 grams per day and contraceptives.

* Subject has a hypersensitivity, intolerance, or contraindication to the use of sumatriptan or naproxen sodium or any of their components or any other 5-HT1 receptor agonist.
* Subject has a history of any gastrointestinal surgery that specifically indicates a past history of bleeding, ulceration or perforation.
* Subject has a history of gastric bypass or stapling surgery.
* Subject has a history of GI ulceration in the past six months or gastrointestinal bleeding in the past year.
* Subject has a history of inflammatory bowel disease.
* Treatment with an investigational drug within 30 preceding the first dose of study medication.
* Positive serum beta-human chorionic gonadotropin test -females.
* Pregnant, actively trying to become pregnant or breast-feeding.
* Subjects with a history of drug or alcohol abuse.
* History of regular alcohol consumption exceeding 7 drinks per week for females or 14 drinks per week for men within 6 months of screening.
* Positive urine drug screen including alcohol at screening.
* Donation of blood in excess of 500 mL within 56 days prior to first dose of study medication.
* Subjects who smoke more than 10 cigarettes per day.
* History of sensitivity to heparin, heparin-induced thrombocytopenia or sensitivity to any of the study medications or components thereof.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05-06 (Actual); Primary Completion 2008-06-14 (Actual); Study Completion 2008-06-14 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) after the second dose and total exposure (measured by AUC(0-∞) calculated as pooled exposure from both the initial and second dose). | ten weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events, blood pressure, pulse, ECGs and clinical laboratory tests. | ten weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Berges A, Walls C, Lener SE, McDonald SA. Pharmacokinetics and tolerability of sumatriptan after single-dose administration of a fixed-dose combination tablet of sumatriptan/naproxen sodium 85/500 mg followed two hours later by subcutaneous sumatriptan 4- or 6-mg injection: a randomized, open-label, three-period crossover study in healthy volunteers. Clin Ther. 2010 Jun;32(6):1165-77. doi: 10.1016/j.clinthera.2010.06.014. PMID 20637969
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 103629 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/103629?search=study&study_ids=103629#rs
- Available data/document: Dataset Specification: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register